CLINICAL TRIAL: NCT06450522
Title: Post-Discharge Pharmacist-led Rapid Medication Optimization for Heart Failure (Post-Discharge PHARM-HF): a Randomized Controlled Trial
Brief Title: Post-Discharge Pharmacist-led Rapid Medication Optimization for Heart Failure (Post-Discharge PHARM-HF)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ricky Turgeon, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H24-00300
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure with Reduced Ejection Fraction HFrEF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacist co-management (Experimental): In addition to usual care, participants with an initial Post-Discharge Medicine Clinic visit randomized to the intervention arm will receive pharmacist co-management of their medications, with the intent of to achieve rapid, maximum-tolerated pharmacotherapy for HF as outlined in the latest guidelines. This intervention will be delivered by a staff pharmacist at the St. Paul's Hospital, using the standard procedures outlined below:
  For HFrEF, where possible, a patient will be prescribed the combination of an ARNI, evidence-based beta-blocker, MRA, and SGLT2i at target HFrEF doses, along with personalized therapies as outlined in the 2021 CCS HF guidelines.
  For HFmrEF, we will target ACEI/ARB/ARNI, beta-blocker, MRA, and SGLT2i. For HFpEF, we will target SGLT2i + MRA +/- ACEI/ARB/ARNI. The intervention will incorporate key components identified in a systematic review of observational studies of pharmacist-led optimization of HF.
  Interventions: Other: Pharmacist co-management of HF medication optimization
- Usual care (Other): Usual care: Both the intervention group and comparator group will receive usual care by the Post-Discharge Medicine Clinic, which does not include clinical pharmacy services. The standard pathway in the St. Paul's Hospital Post-Discharge Medicine Clinic consists of an initial consultation with the clinic internist within 2 weeks of discharge, followed by two visits approximately 1 week apart with the Post-Discharge Medicine Clinic internist, followed by discharge from the clinic.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pharmacist co-management of HF medication optimization — In addition to usual care, participants with an initial Post-Discharge Medicine Clinic visit randomized to the intervention arm will receive pharmacist co-management of their medications, with the intent of to achieve rapid, maximum-tolerated pharmacotherapy for HFrEF as outlined by the 2021 CCS HF guidelines, and for HFmrEF/HFpEF as outlined by the 2022 ACC/AHA HF guidelines. This intervention will be delivered by a staff pharmacist at the St. Paul's Hospital, using the standard procedures outlined below:
  For HFrEF: Where possible, a patient will be prescribed the combination of an ARNI, evidence-based beta-blocker, MRA, and SGLT2i at target HFrEF doses, along with personalized therapies as outlined in the 2021 CCS HF guidelines.
  For HFmrEF: We will target ACEI/ARB/ARNI+BB+MRA+SGLT2i. For HFpEF: We will target SGLT2i+MRA +/- ACEI/ARB/ARNI. The intervention will incorporate key components identified in a systematic review of observational studies of pharmacist-led optimization of HF.
  Arms: Pharmacist co-management
Other: Usual care — Usual care
  Arms: Usual care

SUMMARY:
This study will recruit 100 patients from a post-discharge medicine clinic to test if the addition of a pharmacist to manage heart failure medications can increase appropriate use of these medications. Participants will be randomly assigned to usual care alone or with the addition of a pharmacist to help manage medications. They will be followed for 3 months by telephone/electronically-administered questionnaires, and 12 months using administrative health records. Outcome data will include information from patients on quality of life, treatment burden, medication adherence, as well as information from their medical record on heart failure events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 years;
2. Attending their initial visit to the PDMC;
3. Diagnosis of HF.

Exclusion Criteria:

* None.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Optimization Potential Score | 3 months
  Score that quantifies guideline-directed medical therapy (GDMT) use in heart failure with reduced ejection fraction. The score ranges from 0 (worst) to 10 (best).
  For HFmrEF, this will be modified to assign equal weight to ACEI/ARB/ARNI (score range 0-8).
  For HFpEF, this will be further modified to assign equal weight to ACEI/ARB/ARNI, and to assign no points for beta-blocker use (score range 0-6).

SECONDARY OUTCOMES:
Composite hierarchical outcome | 3 months
  Hierarchical composite outcome of time to all-cause death, time to first all-cause hospitalization, the number of HF events (including HF hospitalizations or emergency department visits for HF), ≥5-point Kansas City Cardiomyopathy Questionnaire-12 summary score improvement, or ≥2-point OPS increase

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No